CLINICAL TRIAL: NCT07330401
Title: Assessment of Cytotoxicity, Genotoxicity in Exfoliated Buccal Mucosa Cells Following Exposure to OPG and CBCT Radiations: A Comparative Study Across Age Groups
Brief Title: Assessment of Cytotoxicity, Genotoxicity
Status: Completed | Type: Observational
Sponsor: Yaxin Wang (Other)
Responsible Party: Sponsor-Investigator, Yaxin Wang, master, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Other Study IDs: Universiti Sains Malaysia wang
Record Dates: First submitted 2025-11-22; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Genotoxicity; Cytotoxicity; Ionizing Radiation Exposure; Dental X-Ray Exposure
Keywords: Buccal Mucosa Cells; Micronucleus Assay; Dental Radiography; Orthopantomogram (OPG); Cone Beam Computed Tomography (CBCT); Low-Dose Ionizing Radiation; Age-Related Radiosensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- OPG,15-25 years old
- CBCT,15-25 years old
- OPG,40-50 years old
- CBCT,40-50 years old

SUMMARY:
Goal:

The goal of this observational study is to evaluate the genotoxic and cytotoxic effects of OPG and CBCT on exfoliated buccal mucosal cells

Main question:

Does CBCT cause greater genotoxic and cytotoxic effects on buccal mucosal cells compared with OPG? Buccal epithelial cells were gently exfoliated from participants scheduled to undergo OPG or CBCT imaging. Samples were collected twice-immediately before exposure and again 10-12 days afterward. All participants provided written informed consent prior to inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

Underwent routine dental imaging using OPG or CBCT (no additional radiation for research purposes).

Age 15-25 years or 40-50 years at the time of enrolment.

Able and willing to provide written informed consent (or consent from a legal guardian for minors).

Agreed to provide pre-exposure and follow-up buccal epithelial cell samples.

Exclusion Criteria:

History of systemic diseases, including but not limited to leukemia, lymphoma, rheumatic disorders, or diabetes mellitus.

Prior exposure to head-and-neck radiotherapy, immunosuppressive drugs, or cytotoxic medications.

Presence of active infectious diseases or acute/chronic inflammatory conditions at the time of enrolment.

Clinically visible oral pathological lesions, including mucosal abnormalities, gingivitis, or periodontitis.

Use of removable intra-oral prostheses or appliances (e.g., dentures, orthodontic appliances).

Engagement in smoking, alcohol consumption, or betel-nut chewing.

Diagnostic or therapeutic X-ray exposure within the preceding 3 months.

Previous or current oral mucosal diseases, including oral lichen planus, recurrent aphthous stomatitis, oral candidiasis, HSV infection, leukoplakia, oropharyngeal carcinoma, mucous membrane pemphigoid, or pemphigus vulgaris.

Presence of persistent local irritants, including ill-fitting dental prostheses, sharp teeth/restorations, chemical irritation (acidic foods, alcohol-based mouthwash), or recurrent thermal injury.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adults aged 15-25 years and 40-50 years undergoing routine dental radiographic examination (OPG or CBCT), with follow-up buccal cell sampling for cytogenetic analysis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Change in micronucleated buccal epithelial cells measured by the Buccal Micronucleus Cytome Assay (MN per 2,000 cells) | 10 ±12 days after exposure
  Micronucleated buccal epithelial cells will be quantified using the Buccal Micronucleus Cytome Assay following Sarto et al. (1987) criteria.
  For each participant, 2,000 exfoliated buccal cells will be evaluated at two time points:
  1. immediately before dental X-ray exposure, and
  2. approximately 10 ± 2 days after exposure.
  The primary analysis will report the change in the number of micronucleated cells per 2,000 cells (post-pre difference).
  Micronuclei are identified based on size, morphology, staining characteristics, and separation from the main nucleus.
  Higher post-pre values indicate greater genotoxic response.

CONTACTS AND LOCATIONS:
Locations (1):
- universiti Sains Malaysia hospital, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No